CLINICAL TRIAL: NCT07135804
Title: A Phase II Prospective, Single-Arm, Multicenter Clinical Study of Iparomlimab and Tuvonralimab Injection in the Treatment of Patients With Previously Untreated Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Iparomlimab and Tuvonralimab Injection for Untreated Locally Advanced Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-I-2025-001
Record Dates: First submitted 2025-07-25; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Nasopharyngeal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Eligible subjects are selected according to the inclusion and exclusion criteria. They will receive 3 courses of Iparomlimab and Tuvonralimab Injection during the induction chemotherapy period, undergo standard concurrent chemoradiotherapy as scheduled, and receive 9 cycles of Iparomlimab and Tuvonralimab Injection (5mg/kg, Q3W) in the adjuvant stage. This will continue until the researcher judges that the subject can no longer benefit, the disease progresses, intolerable toxicity occurs, the researcher decides to stop, the subject withdraws informed consent, or death occurs.
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection — Patients will receive Iparomlimab and Tuvonralimab Injection on the basis of 3 cycles of induction chemotherapy, followed by standard concurrent chemoradiotherapy, and then 9 cycles of Iparomlimab and Tuvonralimab Injection as adjuvant therapy
  Other Names: QL1706

SUMMARY:
This is a prospective, multicenter phase II clinical study. The subjects are patients with previously untreated locally advanced nasopharyngeal carcinoma, with clinical staging of IVA, T1-4, N3, M0. The study aims to preliminarily evaluate the efficacy and safety of Iparomlimab and Tuvonralimab Injectionin the treatment of these patients.

DETAILED DESCRIPTION:
Research Objective: To preliminarily evaluate the efficacy and safety of Iparomlimab and Tuvonralimab Injection in the treatment of previously untreated locally advanced nasopharyngeal carcinoma patients.

Study Design: Prospective, multicenter phase II clinical study. Study Subjects: Previously untreated locally advanced nasopharyngeal carcinoma patients with clinical stage: IVA, T1-4, N3, M0.

Sample Size: It is assumed that the 3-year distant metastasis free survival (DMFS) rate of T1-4N3M0 nasopharyngeal carcinoma patients after standard treatment is 74%, and the 3-year DMFS rate after combining with Iparomlimab and Tuvonralimab Injection in the induction and adjuvant stages for T1-4N3M0 nasopharyngeal carcinoma patients is 90%. With a two-sided α=0.05 and power of 80%, and considering a 10% dropout rate, the total sample size is calculated to be 45 cases.

Inclusion Criteria: Refer to the corresponding section. Exclusion Criteria: Refer to the corresponding section. Treatment Plan: Eligible subjects are selected according to the inclusion and exclusion criteria. They will receive 3 courses of Iparomlimab and Tuvonralimab Injection during the induction chemotherapy period, undergo standard concurrent chemoradiotherapy as scheduled, and receive 9 cycles of Iparomlimab and Tuvonralimab Injection (5mg/kg, Q3W) in the adjuvant stage. This will continue until the researcher judges that the subject can no longer benefit, the disease progresses, intolerable toxicity occurs, the researcher decides to stop, the subject withdraws informed consent, or death occurs.

Study Endpoints:

Primary Study Endpoint: 3-year distant metastasis-free survival (DMFS). Secondary Study Endpoints: Objective response rate (ORR), disease control rate (DCR), duration of response (DoR), progression-free survival (PFS), overall survival (OS), safety and tolerability (according to CTCAE 5.0 criteria).

Exploratory Endpoints: Analysis of the correlation between PD-L1 expression and CTLA-4 expression in tumor tissues and the anti-tumor activity of Iparomlimab and Tuvonralimab Injection, and the correlation between EBV-DNA quantification and prognosis.

Statistical Analysis Methods: The chi-square test will be used for comparing rates. Time-event data will be used to estimate the survival function by the Kaplan-Meier method, draw survival curves, and estimate the median time and its 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Have fully understood the study and voluntarily signed the informed consent form
* Newly diagnosed and histologically confirmed nasopharyngeal non-keratinizing carcinoma (T1-4, N3, M0, Stage IVA) with no evidence of distant metastatic disease
* Induction chemotherapy regimen: gemcitabine plus cisplatin; radiotherapy prescription dose is 70Gy, with 32-35 fractions, single dose of 2.0-2.2Gy, to be completed within 7 weeks (once a day, 5 times a week); concurrent cisplatin 80mg/m² during radiotherapy
* According to Response Evaluation Criteria in Solid Tumors (RECIST 1.1), have at least one measurable lesion (except for brain metastases)
* ECOG performance status of 0-1
* Male or female patients aged 18-70 years
* Estimated survival time ≥ 3 months
* Laboratory test values within 7 days before enrollment must meet the following standards (no blood components, cell growth factors, albumin or other corrective treatment drugs are allowed within 14 days before obtaining laboratory tests):

  1. Absolute neutrophil count (ANC) ≥ 1.5×10⁹ /L;
  2. Platelets ≥ 100×10⁹ /L;
  3. Hemoglobin ≥ 9g/dL;
  4. Serum albumin ≥ 2.8g/dL;
  5. Total bilirubin ≤ 1.5×ULN, ALT, AST and/or AKP ≤ 2.5×ULN; if there is liver metastasis, ALT and/or AST ≤ 5×ULN; if there is liver metastasis or bone metastasis, AKP ≤ 5×ULN;
  6. Serum creatinine ≤ 1.5×ULN or creatinine clearance rate > 60 mL/min (Cockcroft-Gault, see Appendix II);
  7. Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤ 1.5×ULN (screening is allowed for those receiving stable doses of anticoagulant therapy such as low molecular weight heparin or warfarin with INR within the expected therapeutic range of anticoagulants)
* Female patients of childbearing age or male patients whose sexual partners are of childbearing age must take effective contraceptive measures throughout the treatment period and within 6 months after the last dose
* Researchers consider that the patient can benefit from the study
* Expected survival time of ≥3 months
* Laboratory test values within 7 days before enrollment must meet the relevant standards (no administration of any blood components, cell growth factors, albumin or other corrective treatment drugs is allowed within 14 days before obtaining the laboratory tests)
* Female patients of childbearing age or male patients whose sexual partners are of childbearing age must use effective contraceptive measures throughout the treatment period and for 6 months after the last dose
* The investigator determines that the patient is likely to benefit from the treatment

Exclusion Criteria:

* Received anti-tumor cytotoxic drug therapy, biological drug therapy (such as monoclonal antibodies), immunotherapy (such as interleukin-2 or interferon), or other investigational drug therapy within 4 weeks before enrollment, except for corticosteroids
* Previously received anti-VEGFR and other vascular-targeted drug therapy
* Judged by the researcher to have impaired immunity
* Underwent major surgical operation within 4 weeks before enrollment or has not fully recovered from previous surgery (the definition of major surgical operation refers to grade 3 and 4 operations specified in the "Administrative Measures for Clinical Application of Medical Technologies" implemented on May 1, 2009)
* Toxic reactions from previous anti-tumor treatment have not recovered to CTCAE grade 0-1, except for the following situations:

  1. Alopecia;
  2. Pigmentation;
  3. Peripheral neurotoxicity has recovered to < CTCAE grade 2;
  4. Long-term toxicity caused by radiotherapy, which cannot recover as judged by the researcher
* Grade 3-4 bleeding or high bleeding risk caused by underlying malignant tumors (such as but not limited to tumors surrounding or infiltrating large blood vessels, i.e., carotid artery, jugular vein) and/or specific other high-risk characteristics (e.g., arteriovenous fistula)
* Previously or currently suffering from other malignant tumors (except for well-controlled non-melanoma skin basal cell carcinoma, breast/cervical carcinoma in situ, and other malignant tumors that have been effectively controlled without treatment in the past five years)
* Subjects with any active autoimmune disease or a history of autoimmune diseases (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or asthma that has been completely relieved in childhood and do not require any intervention in adulthood can be included; those with asthma requiring medical intervention with bronchodilators cannot be included)
* Previously used anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, or anti-CTLA-4 antibody (or any other antibody acting on T cell co-stimulation or checkpoint pathways)
* Subjects with active pulmonary tuberculosis (TB) who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year before screening
* Received any anti-infective vaccine (such as influenza vaccine, varicella vaccine, etc.) within 4 weeks before enrollment
* Pregnant or lactating women
* HIV positive
* Patients with acute or chronic active hepatitis B or C infection, with hepatitis B virus (HBV) DNA > 2000 IU/ml or 10⁴ copies/ml, hepatitis C virus (HCV) RNA > 10³ copies/ml; simultaneous positivity for hepatitis B surface antigen (HbsAg) and anti-HCV antibody. Those who are below the above standards after nucleotide antiviral treatment can be enrolled
* Any life-threatening bleeding event within the previous 3 months, including those requiring blood transfusion, surgery or local treatment, and continuous drug treatment
* A history of arterial or venous thromboembolic events within the previous 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or any other serious thromboembolic history. Except for those with implantable venous access port or catheter-derived thrombosis, or superficial venous thrombosis, whose thrombosis is stable after conventional anticoagulant therapy. Prophylactic use of low-dose low molecular weight heparin (such as enoxaparin 40mg/day) is allowed
* Uncontrolled hypertension, with systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg after optimal medical treatment, or a history of hypertensive crisis or hypertensive encephalopathy
* Used aspirin (> 325mg/day) or other drugs known to inhibit platelet function such as dipyridamole or clopidogrel for 10 consecutive days within 2 weeks before the first dose
* Symptomatic congestive heart failure (New York Heart Association class II-IV). Symptomatic or poorly controlled arrhythmias. A history of congenital long QT syndrome or corrected QTc > 500ms at screening (calculated using the Fridericia method)
* Severe bleeding tendency or coagulation dysfunction, or receiving thrombolytic therapy
* A history of gastrointestinal perforation and/or fistula within the previous 6 months, a history of intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive intestinal resection (partial colon resection or extensive small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or long-term chronic diarrhea
* Known allergy to any component of PD-1 and CTLA-4 antibodies; or have had a severe allergic reaction to other monoclonal antibodies in the past
* Any other clinically significant diseases or conditions that the researcher believes may affect protocol compliance, or affect the subject's signing of the informed consent form (ICF), or make them unsuitable for participating in this clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
3-year distant metastasis-free survival (DMFS) as assessed by imaging examinations (including CT, MRI, PET-CT) and clinical evaluations to determine the time from randomization to the first occurrence of distant metastasis or death from any cause | Up to 3 years after enrollment (each follow-up cycle is 3 months for the first two years, 6 months for the third year)
  DMFS will be calculated as the time from the date of enrollment to the date of first documented distant metastasis (confirmed by imaging modalities such as CT, MRI, or PET-CT) or death from any cause, whichever occurs earlier. Patients who are lost to follow-up or withdraw from the study will be censored at the last date they were known to be free of distant metastasis and alive. The 3-year DMFS rate will be estimated using the Kaplan-Meier method, with the 95% confidence interval reported.
Objective response rate (ORR) of the tumor as assessed by RECIST 1.1 criteria, including complete response (CR) and partial response (PR) confirmed by imaging examinations (CT, MRI) | Every 9 weeks during treatment (each treatment cycle is 3 weeks) and at the end of treatment
  ORR is defined as the proportion of participants with best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1. CR is defined as the disappearance of all target lesions and no new lesions, with normalization of tumor marker levels if applicable. PR is defined as at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum of longest diameters. Responses must be confirmed by a subsequent assessment at least 4 weeks after the initial documentation of CR or PR